CLINICAL TRIAL: NCT06883539
Title: A Phase I Open-label Dose-finding Study to Assess the Safety, Tolerability, Pharmacokinetics and Efficacy of LXP1788 Injection in Patients with Advanced Solid Tumors.
Brief Title: A Phase I Study of LXP1788 Injection with Advanced Solid Tumors.
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: LaunXP Biomedical Co., Ltd. (Industry)
Collaborators: Efficient Pharma Management Corp. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DBPR114-101
Record Dates: First submitted 2025-03-06; First posted 2025-03-19 (Actual); Last update posted 2025-03-19 (Actual); Status verified 2025-03

CONDITIONS: Solid Tumor Malignancies, Cancer; Solid Cancers; Solid Tumor Cancer; Solid Tumor, Unspecified, Adult; Solid Tumour; Solid Tumors Refractory to Standard Therapy; HCC - Hepatocellular Carcinoma; RCC, Renal Cell Cancer; Pancreas Cancer
Keywords: Phase 1; LXP1788; LAUNXP; DBPR114-101; solid tumor; cancer; Hepatocellular carcinoma; Pancrease Cancer; Renal Cell Carcinoma; Tyrosine kinase inhibitor
MeSH Terms: conditions — Neoplasms; Carcinoma, Hepatocellular; Carcinoma, Renal Cell; Pancreatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- LXP1788 Injection will be administered intravenously once a week in a 28-day treatment cycle. (Experimental)
  Interventions: Drug: LXP1788 is administered intravenously via Port-A

INTERVENTIONS:
Drug: LXP1788 is administered intravenously via Port-A — LXP1788 Injection is formulated as a solution for injection and will be administered intravenously for 60 minutes on days 1, 8, 15, 22 of the cycle. Each cycle will be 28 days.

SUMMARY:
A Phase I, open-label, first-in-human study to determine the MTD, recommended phase 2 dose (RP2D), assess the safety, tolerability, pharmacokinetics and preliminary anti-tumor activity of LXP1788 Injection in patients with advanced solid tumor.

Patients with advanced solid tumors that are refractory to currently available therapies or for whom no effective treatment is available will be selected.

The main questions it aims to answer are:

1. To determine the maximum tolerated dose (MTD) and the recommended phase 2 dose (RP2D) of LXP1788 Injection
2. To evaluate the pharmacokinetics (PK) of LXP1788 Injection

ELIGIBILITY:
Inclusion Criteria:

1. Written (signed) Informed Consent.
2. Male or female ≥ 18 years old.
3. Life expectancy > 8 weeks.
4. Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
5. A histologically or cytologically confirmed, advanced solid tumor that is refractory to currently available therapies or for which no effective treatment is available.
6. Measurable disease per RECIST 1.1.
7. Willing to have a tumor biopsy or having tissue sample from a previous biopsy available in the tissue bank for analysis that had been collected in the past 3 years.

Exclusion Criteria:

1. Significant concurrent medical diseases, such as congestive heart failure, unstable angina, acute or recent myocardial infarction (< 6 months before enrollment), COPD with frequent exacerbations, uncontrolled hypertension (systemic blood pressure >= 160 mmHg and/or diastolic blood pressure >= 100 mmHg with or without anti-hypertensive medication), recent CVA (< 6 months before enrollment), or active infection which requires treatment withintravenous antibiotics.
2. Patients with symptomatic CNS metastases who are neurologically unstable, receiving radiotherapy for the CNS lesion, or requiring increasing dose of steroids to control their CNS disease.

   Asymptomatic patients with metastatic brain disease who have been on a stable dose of steroids for less than 14 days prior to screening.
3. Inadequate bone marrow reserve or organ function as demonstrated by any of the following laboratory values:

   Bone marrow:
   * Absolute neutrophil count (ANC) < 1.5 x 10^9/L
   * Platelet count < 100 x 10^9/L
   * Hemoglobin < 9 g/dL
   * Having had a blood transfusion within 2 weeks of screening date is also not allowed.

   Hepatic:
   * Total bilirubin > 1.5 x ULN
   * AST and ALT > 3 x ULN if no liver metastases
   * AST and ALT > 5 x ULN in the presence of liver metastases

   Renal:

   ⚫ Estimated creatinine clearance (CrCL) < 60 mL/min per the Cockcroft and Gault formula
4. Known history of human immunodeficiency virus (HIV)-1 or -2 infection.
5. Psychiatric disorders that would compromise the patient's compliance or ability to give consent.
6. Major surgical intervention within 4 weeks of the first dose of LXP1788 Injection or with ongoing postoperative complications.
7. Toxicities from any prior therapy, surgery, or radiotherapy that did not resolve to grade 0 or 1 as per the National Cancer Institute (NCI) - Common Terminology Criteria for Adverse Events (CTCAE) Version 5.0, with the exception of alopecia, skin hyperpigmentation or hypopigmentation.
8. Underlying medical conditions that, in the investigator's opinion, will make the administration of LXP1788 Injection hazardous or obscure the interpretation of toxicities or adverse events.
9. Exposure to any other investigational or commercial anti-cancer agents or curative therapies within 28 days or 5 half-lives (whichever is shorter), before the first dose of LXP1788 Injection. Exposure to radiation therapy for non-curative purposes or pain control may be permitted under the judgement of the investigator.
10. Judgment by the investigator that the patient should not participate in the study because the patient is unlikely to comply with study procedures, restrictions, or requirements.
11. Pregnancy or breast feeding.
12. Women or men of childbearing potential not willing to use effective means of contraception.
13. Positive test for hepatitis B (HBsAg) or hepatitis C (positive HCV antibody with detectable HCV RNA).
14. History of allergic reactions to any component of LXP1788 Injection.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2024-12-31 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2028-06-30 (Estimated)

PRIMARY OUTCOMES:
To determine the MTD and potential phase 2 dose regimen(s) of LXP1788 Injection | 2 years
To characterize the plasma PK profile of LXP1788 following IV administration of LXP1788 Injection | 2 years
  PK blood samples to determine plasma concentrations of LXP1788 will be collected at the time points listed in the schedule of events table. Where possible, the plasma concentration-time data will be used to calculate the following parameters for LXP1788 Injection by non-compartmental methods: Maximum plasma concentration (Cmax), dose-normalized Cmax (Cmax/D), area under the concentration-time curve from time 0 to 24 hours post-dose (AUC0-24), dose-normalized AUC0-24 (AUC0-24/D), AUC from time 0 to the last quantifiable concentration (AUC0-last), dose-normalized AUC0-last (AUC0-last/D), AUC from time 0 extrapolated to infinity (AUC0-inf), dose-normalized AUC0-inf (AUC0-inf/D), time to Cmax (tmax), plasma clearance (CL), volume of distribution (Vz), terminal rate constant (λz), and terminal elimination half-life (t1/2).

SECONDARY OUTCOMES:
To assess the safety, tolerability, and dose-limiting toxicity (DLT) of LXP1788 Injection | 2 years
  To assess the safety, tolerability, and dose-limiting toxicity (DLT) of LXP1788 Injection
To assess exposure levels to LXP1788 | 2 years
  To assess exposure levels to LXP1788
To assess anti-tumor activity of LXP1788 Injection | 2 years
  To assess anti-tumor activity of LXP1788 Injection
  * Objective response rate (ORR) using RECIST 1.1 for solid tumor
  * Time to tumor progression (TTP)
  * Disease control rate (DCR)
  * Clinical benefit rate (CBR)
  * Duration of response (DoR)
  * Progression free survival (PFS)

CONTACTS AND LOCATIONS:
Locations (2):
- Taiwan (2):
  - China Medical University Hospital, Taichung
  - National Cheng Kung University Hospital, Tainan

IPD SHARING:
Plan to Share IPD: No